CLINICAL TRIAL: NCT02452801
Title: A Phase 1 Study of the Pharmacokinetics, Safety, and Tolerability of ALKS 5461 in Subjects With Hepatic Impairment
Brief Title: Pharmacokinetics and Safety of ALKS 5461 in Healthy Subjects and Subjects With Hepatic Impairment and Normal Hepatic Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alkermes, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALK5461-215
Record Dates: First submitted 2015-05-21; First posted 2015-05-25 (Estimated); Last update posted 2016-02-04 (Estimated); Status verified 2016-02

CONDITIONS: Hepatic Impairment
MeSH Terms: interventions — ALKS 5461

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ALKS 5461 (Experimental): Sublingual tablet
  Interventions: Drug: ALKS 5461

INTERVENTIONS:
Drug: ALKS 5461 — Single dose, given orally

SUMMARY:
This study will evaluate the effect of various degrees of hepatic function on the pharmacokinetics and safety of ALKS 5461.

ELIGIBILITY:
Inclusion Criteria:

For all subjects:

* Has a body mass index (BMI) of 18.0-35.0 kg/m2 and a total body weight >50 kg
* Agrees to use an approved method of contraception for the duration of the study
* Additional criteria may apply

For subjects with hepatic impairment:

* Has mild, moderate, or severe hepatic impairment
* Has hepatic dysfunction due to hepatocellular disease
* Additional criteria may apply

Exclusion Criteria:

For all subjects:

* Has any past history or current finding of a clinically significant observed abnormality, psychiatric or medical condition other than hepatic impairment
* Has a history of gastrointestinal surgery, excluding appendectomy or cholecystectomy
* Is pregnant, planning to become pregnant, or lactating
* Has a history of clinically significant allergy or a hypersensitivity to opioids
* Additional criteria may apply

For subjects with hepatic impairment:

* Has evidence of hepatocellular carcinoma, acute liver disease, biliary obstruction, severe ascites, severe portal hypertension, surgical systemic shunts, or other clinically relevant liver-related disorder or condition
* Has received a liver transplant
* Has had esophageal variceal bleeding in the past 2 months
* Additional criteria may apply

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-05; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time curve from time 0 to infinity (AUC0-inf) following a single dose of ALKS 5461 | Up to 168 hours postdose
Area under the plasma concentration versus time curve from time 0 to time of last measureable concentration (AUC0-last) following a single dose of ALKS 5461 | Up to 168 hours postdose
Maximum observed plasma concentration (CMAX) following a single dose of ALKS 5461 | Up to 168 hours postdose

SECONDARY OUTCOMES:
Time to reach maximum plasma concentration (TMAX) | Up to 168 hours postdose
Terminal elimination half-life (T1/2) | Up to 168 hours postdose
Apparent clearance (CL/F) | Up to 168 hours postdose
Apparent volume of distribution (Vz/F) | Up to 168 hours postdose
Incidence of adverse events (AEs) | Up to 14 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sanjeev Pathak, MD, Study Director — Alkermes, Inc.
Locations (1):
- Alkermes Investigational Site, Orlando, Florida, United States